CLINICAL TRIAL: NCT05234879
Title: The Feasibility of Frame Running as an Exercise Option for People With Multiple Sclerosis With Impaired Balance and Mobility
Brief Title: The Feasibility of Frame Running as an Exercise Option for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Collaborators: Multiple Sclerosis Society of Great Britain (Unknown)
Responsible Party: Principal Investigator, Marietta van der Linden, Senior research fellow, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PM1951QMU
Record Dates: First submitted 2022-01-20; First posted 2022-02-10 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frame Running intervention (Experimental): Participants will be invited to 12 Frame Running training sessions
  Interventions: Other: Frame Running

INTERVENTIONS:
Other: Frame Running — Frame Running (FR) provides an opportunity for people with walking and balance problems to walk or run safely without the risk of falling. The frame consists of three wheels and has a saddle and handlebars like a trike without pedals.

SUMMARY:
There is ample evidence that regular exercise can reduce MS specific symptoms and improve health and wellbeing in people with MS. However, for people with MS to engage in exercise activities long term, it is important that they are offered a range of exercise opportunities that are safe, feasible and potentially effective to reduce MS symptom. This will allow people to select an activity they enjoy, is adapted to their needs and thus are more sustainable long-term. Frame Running (FR) provides an opportunity for people with walking and balance problems to walk or run safely without the risk of falling. The frame consists of three wheels and has a saddle and handlebars like a trike without pedals. The proposed mixed methods study aims to examine the feasibility and acceptability of FR as a sustainable aerobic exercise option for people with MS and the feasibility of conducting a future definite trial into the impact of FR on functional mobility, fatigue, cardiorespiratory function and psychosocial outcomes. People who experience problems with their walking and/or balance will be eligible to take part in this study which consists of a 12 weekly group FR training sessions led by a qualified coach. FR training attendance, recruitment, retention, outcome measure completion and adverse events will be recorded and the participant views on the feasibility, acceptability and impact of FR will be explored through the use of focus groups. Physical function, physical activity and psychosocial outcomes will be assessed at baseline, 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* People with a definite diagnosis of MS according to the revised MacDonald criteria, aged 18 and over, experiencing walking or balance difficulties but able to transfer independently will be eligible to take part in this study. This equates to people with an EDSS of 3.5 to 7. In order to be eligible for taking part in the Frame Running sessions, people should also be able comprehend and follow instructions relating to participation training as well as have sufficient understanding of the English language to complete the consent forms and questionnaires

Exclusion Criteria:

* Those with contraindications to exercise, those unable to safely propel the frame for any distance on their own using the try-out sessions and those with more than 10 hours of FR experience will be excluded from participation in this study. Other exclusion criteria are lower limb surgery less than 3 months prior to the start of the study, having started disease modifying and/or spasticity treatment less than 3 months prior to the start of the study and severe visual impairment affecting the ability to safely take part in Frame Running training sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Exercise Self Efficacy Scale | baseline
  questionnaire (range 10-40) higher scores indicate higher self-efficacy
Exercise Self Efficacy Scale | 12 weeks
  questionnaire (range 10-40) higher scores indicate higher self-efficacy
Psychological Impact of Assistive Devices Scale | baseline
  questionnaire (range -3 to 3) higher score indicate improvement in psychosocial impact
Psychological Impact of Assistive Devices Scale | 12 weeks
  questionnaire (range -3 to 3) higher score indicate improvement in psychosocial impact
Five times sit-to-stand test | baseline
  measurer of functional strength, Duration, measured in seconds
Five times sit-to-stand test | 12 weeks
  measurer of functional strength, Duration, measured in seconds
Canadian Occupational Performance Measure | baseline
  semi-structured interview (ratings range from 1 to 10, higher scores indicate higher perceived improvement in function
Canadian Occupational Performance Measure | 12 weeks
  semi-structured interview (ratings range from 1 to 10, higher scores indicate higher perceived improvement in function
Resting blood pressure | baseline
  resting blood pressure in mmHg
Resting blood pressure | 12 weeks
  resting blood pressure in mmHg
six minute Frame Running test | baseline
  measured in meters travelled during 6 minutes, test conducted on a running track
six minute Frame Running test | 11 weeks
  measured in meters travelled during 6 minutes, test conducted on a running track
Frame Running shuttle run/walk test | baseline
  test conducting on the running track, outcome is number of shuttles performed
Frame Running shuttle run/walk test | 12 weeks
  test conducting on the running track, outcome is number of shuttles performed
weekly step count | baseline
  Measured using an ActivPAL activity monitor
weekly step count | 11 weeks
  Measured using an ActivPAL activity monitor
Fatigue Scale for Motor and Cognitive Functions (FSMC) | baseline
  questionnaire (range 20 to 100) higher scores indicate higher self-reported fatigue
Fatigue Scale for Motor and Cognitive Functions (FSMC) | 12 weeks
  questionnaire (range 20 to 100) higher scores indicate higher self-reported fatigue
Multiple Sclerosis Walking Scale | baseline
  questionnaire (range 12-60) higher scores indicate higher self-reported limitation in walking ability
Multiple Sclerosis Walking Scale | 12 weeks
  questionnaire (range 12-60) higher scores indicate higher self-reported limitation in walking ability
Godin Leisure time exercise questionnaire | baseline
  questionnaire (range 0-119) higher scores indicate higher level of leisure time exercise participation
Godin Leisure time exercise questionnaire | 12 weeks
  questionnaire (range 0-119) higher scores indicate higher level of leisure time exercise participation

SECONDARY OUTCOMES:
number of weekly training session attended | 12 weeks
  range 0 to 12
Heart rate during the training session | 3 weeks
  maximum HR and time spent in HR zones
Heart rate during the training session | 8 weeks
  maximum HR and time spent in HR zones

OTHER OUTCOMES:
focus groups | 12 weeks
  insights into participant's views on positive and negative experiences or impacts and thoughts on ongoing participation

CONTACTS AND LOCATIONS:
Overall Officials: Marietta L van der Linden, PhD, Principal Investigator — Queen Margaret University
Locations (1):
- Queen Margaret University, Musselburgh, East Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
overall study outcomes will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available as part of a publication which expected to be 31/12/2023 the latest